CLINICAL TRIAL: NCT00034502
Title: A Trial of ALIMTA (Pemetrexed) Plus Irinotecan in Patients Who Have Been Previously Treated For Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 2927; H3E-MC-JMDO
Record Dates: First submitted 2002-04-29; First posted 2002-04-30 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; Irinotecan

INTERVENTIONS:
Drug: ALIMTA
Drug: irinotecan

SUMMARY:
This is a non-randomized study in patients who have received prior 5-FU therapy for colorectal cancer. The objective of this trial is to establish a maximum tolerated dose of ALIMTA and irinotecan given in combination as well as to assess the safety and efficacy of this combination for patients with locally advanced or metastatic colorectal cancer. ALIMTA and irinotecan will be given every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of locally or metastatic colorectal cancer
* Prior therapy with 5-FU for metastatic cancer
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Inability to interrupt aspirin therapy
* Brain metastasis
* Patients who have been treated previously with ALIMTA or irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Pittsburgh, Pennsylvania
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Bielefeld, North Rhine-Westphalia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Homburg/Saar
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., München